CLINICAL TRIAL: NCT01058473
Title: Psychometric Evaluation of the Inpatient Pediatric Physical Activity Questionnaire (IPPAQ) in Pediatric Patients With Sickle Cell Disease Hospitalized With Vasoocclusive Pain
Brief Title: Psychometric Evaluation of the IPPAQ in Pediatric Patients With Sickle Cell Disease Hospitalized With Vasoocclusive Pain
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, William Zempsky, MD, Director, Pain Relief Program, Connecticut Children's Medical Center
Other Study IDs: CCMC IRB Number 09-115
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Sickle Cell Disease; Pain
Keywords: Sickle Cell Disease; Pain; Assessment
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sickle Cell Disease

SUMMARY:
Historically, sickle cell disease has not been viewed in the chronic pain paradigm because of its recurrent nature. Patients with sickle cell disease may be hospitalized for extended periods of time. As the hospital stay progresses, patients with SCD pain are often observed by clinicians to have improvements in function in areas such as self-care, mobility, and recreation despite continued self-report of high pain scores. This pattern of functional improvement with continued report of high pain intensity scores is common in patients with recurrent and chronic pain. A functional assessment tool that can assess function in the acute inpatient setting is needed.

The purpose of this study is to evaluate the Inpatient Pediatric Physical Activity Questionnaire (IPPAQ), as a measure of daily function in children with sickle cell disease hospitalized with vasoocclusive pain.

DETAILED DESCRIPTION:
Refer to Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Documented sickle cell disease
* Sudden onset of pain consistent with vasoocclusive episode at the time of hospitalization.
* Pain requiring hospitalization and placement on standard clinical guideline for management of acute pain in sickle cell disease during hospitalization
* Cognitive ability to report pain on a 0-10 Numerical Rating Scale (NRS)
* Parental/patient consent and child assent

Exclusion Criteria:

* Primary diagnosis other than vasoocclusive pain
* Concurrent Acute Chest Syndrome (ACS)
* Patient previously enrolled in this study
* Inability to understand English

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults with sickle cell disease.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
IPPAQ | 1 day
  This is a functional assessment tool for pediatric sickle cell patients that is admisistered once a day.

CONTACTS AND LOCATIONS:
Overall Officials: William T. Zempsky, M.D., Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States